CLINICAL TRIAL: NCT05961254
Title: Role of Airwayultrasound in Predicting Difficult Endotracheal Intubation in Patients Undergoing General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Meril Nassry Saleeb, Resident-Anesthesia,ICU and Pain management department-sohag hospital university, Sohag University
Other Study IDs: Soh-Med-23-07-19MS
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Predict Diificult Endotracheal Intubation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: assesment of difficult endotracheal intubation by airway ultrasound — preoperative assesment of airway by ultrasound to predict difficult endotracheal intubation in patients undergoing general anesthsia

SUMMARY:
Unpredictable difficult endotracheal intubation remains a challenge especially if difficult ventilation occurs. Difficult intubation is associated with many severe fatal complications including air way trauma, laryngospasm, hypoxemia, arrhythmias and potential cardiac arrest. Therefore, preoperative evaluation and prediction of potential difficult airway is very important.

Several screening tests are used in clinical practice to identify patients at the risk of difficult airway. Despite their accuracy and beneﬁt, a small number of patients classiﬁed to an easy airway may still present an unexpected difficulty. Predicting a difficult airway is not at all an easy task for all patients .

Incidence of difficult airway and difficult intubation varies from 5% to 22% with important implications for clinical practice and patients' outcomes .

There are multiple scores used for airway assesment ,the commonest one is LEMON score. LEMON is an airway assessment score that measures factors associated with difficult intubation such as obesity, head and neck movement, jaw movement , receding mandible, long upper incisors, Mallampatti scores, maxillary incisor characteristics, decreased mouth opening ,shorten thyromental distance and short neck .

Diagnostic criteria for LEMON scoring system :

L- Look. E- Evaluation using the 3-3-2 rule. M- Mallampati. O- Obstruction. N- Neck mobility. Ultrasound (US) imaging technique is simple, portable, noninvasive tool helpful for airway assessment and management. In the last few years, there have been some reports that described various roles of US imaging in airway management. It helps in rapid assessment of the airway anatomy, not only in operation theatre but also in the intensive care unit and emergency department.

Various clinical applications of US imaging of the upper airway include identification of endotracheal tube (ETT) placement, guidance of percutaneous tracheostomy and cricothyroidotomy, detection of subglottic stenosis, prediction of difficult intubation and post-extubation stridor, prediction of paediatric ETT and double-lumen tube (DLT) size.

Recently there are researches about airway assesment by ultrasound. Several airway assesment indicies are used to help in prediction of difficult endotracheal intubation. The most commonly used indices are distance from skin to epiglottis, distance from skin to vocal cord level, and distance from skin to hyoid bone.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients from 18- 50 yrs old
* Patients who require endotracheal intubation for surgery under general anesthesia.

Exclusion Criteria:

* Patients with history of previous difficult intubation.
* Neck deformity such as swelling , scar ,etc.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients from 18- 50 yrs old Patients who require endotracheal intubation for surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
ultasound airway assesment index ..distance from skin to epiglottis | 6 months
  to measure distance from skin to epiglottis
ultasound airway assesment index ..distance from skin to hyoid bone | 6 months
  to measure distance from skin to hyoid bone
ultasound airway assesment index ..distance from skin to vocal cord | 6 months
  to measure distance from skin to vocal cord

SECONDARY OUTCOMES:
airway ultrasound and LEMON score | 6 months
  compare between LEMON score and airway ultrasound in predicting difficult airway.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roth D, Pace NL, Lee A, Hovhannisyan K, Warenits AM, Arrich J, Herkner H. Bedside tests for predicting difficult airways: an abridged Cochrane diagnostic test accuracy systematic review. Anaesthesia. 2019 Jul;74(7):915-928. doi: 10.1111/anae.14608. Epub 2019 Mar 6. PMID 30843190
- [Background] Detsky ME, Jivraj N, Adhikari NK, Friedrich JO, Pinto R, Simel DL, Wijeysundera DN, Scales DC. Will This Patient Be Difficult to Intubate?: The Rational Clinical Examination Systematic Review. JAMA. 2019 Feb 5;321(5):493-503. doi: 10.1001/jama.2018.21413. PMID 30721300
- [Background] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488
- [Background] Frerk C, Mitchell VS, McNarry AF, Mendonca C, Bhagrath R, Patel A, O'Sullivan EP, Woodall NM, Ahmad I; Difficult Airway Society intubation guidelines working group. Difficult Airway Society 2015 guidelines for management of unanticipated difficult intubation in adults. Br J Anaesth. 2015 Dec;115(6):827-48. doi: 10.1093/bja/aev371. Epub 2015 Nov 10. PMID 26556848